CLINICAL TRIAL: NCT04714788
Title: A Mobile App to Improve Participation in Following-up Cohorts of Individuals Born Preterm: a Pragmatic Multicenter Randomized Controlled Trial
Brief Title: A Mobile App to Improve Participation in Following-up Cohorts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Saude Publica da Universidade do Porto (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Netherlands Organisation for Scientific Research (Other Government); University of Tartu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CE20160
Record Dates: First submitted 2021-01-08; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Participants of Longitudinal Cohort Studies; Controls
Keywords: Cohort Studies; Mobile Applications; Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group RECAP_MyLife mobile app (Experimental): Participants in the intervention group will be instructed to use the mobile app daily for four weeks.
  Interventions: Device: RECAP_MyLife mobile app
- Control group (Active Comparator): Comparator will be the usual data collection method applied by the cohorts.
  Interventions: Other: Usual data collection methods

INTERVENTIONS:
Device: RECAP_MyLife mobile app — The intervention will be the use of a mobile application for collecting data from cohorts participants, envisioning to engage participants and collect continuous unbiased records. Participants in the intervention group will install the mobile application on their smartphones on the beginning of the trial and will be asked to self-report information on mood every day. Simultaneously, physical activity (number of steps) will be passively tracked through real-time information.
  Participants will complete baseline and post-intervention measures of mood status based on the "Circumplex Mood Model" and IPAQ-Short form. Following these measures, participants will be asked to complete questionnaires on usability (SUS scale) and acceptability of the intervention.
  Arms: Intervention group RECAP_MyLife mobile app
Other: Usual data collection methods — Participants in this group will provide data through usual types of data collection methods (face-to-face assessments, mailed questionnaires, online questionnaires).
  Arms: Control group

SUMMARY:
The main objective is to test the superiority of a newly developed mobile application - RECAP_MyLife - for data collection in cohort studies in order to increase participation in follow-up evaluations. We hypothesize that data collection through a mobile app will contribute to improvements in participation.

An accurate assessment of the potential benefits and drawbacks of using this mobile technology tool for data collection in cohort studies will be conducted. For such, the study will be conducted in three cohorts developed in different temporal, cultural, and geographic contexts, increasing the generalization of the results found. This evaluation is intended to contribute to the development of more appropriate tools for data collection and consequently to increase participation in epidemiological studies.

DETAILED DESCRIPTION:
This is a multicenter, two-arm, parallel unmasked pragmatic randomized controlled trial with baseline and post-intervention (4 weeks from baseline) assessments. A convenience sample of participants of three population-based cohorts of individuals born very preterm and/or very low birth weight will be randomized and allocated 1:1 to either a mobile app intervention group or into the control arm (usual data collection methods).

Secondary aims of this study are:

1. To evaluate the usability and acceptability of the mobile app among cohort participants.
2. To investigate the potential Hawthorne effect on the results on physical activity behavior and mood status.
3. To measure the agreement between passively tracked physical activity by the mobile app and physical activity measured weekly with a self-reported questionnaire.
4. To measure the agreement between mood status collected by the mobile app through Ecological Momentary Assessment and mood status measured weekly with a self-reported questionnaire.
5. To survey participant's preferences about the different data collection methods.

Intention-to-treat approach will be applied in the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 16 years or over
* Individuals with no evidence of visual impairment, physical condition that may affect the ability to walk, or major cognitive or motor disabilities until the enrollment of the study
* Individuals owning a smartphone with an Android software version 7 or newer.

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Participation | Baseline
  Defined as the total number of individuals who give consent to participate divided by the number of eligible individuals invited for the study.

SECONDARY OUTCOMES:
Completion rates | 4- weeks
  Defined as the total number of participants who complete the follow-up evaluation divided by the number of participants who initiated the trial.
Usability | 4-weeks
  System Usability Scale (SUS)
Acceptability | 4- weeks
  Post-intervention questionnaire
Hawthorne effect - Physical activity | 1-week
  It will be measure if the data collection method affects physical activity, by comparing physical activity behavior (IPAQ-S) at baseline with results collected over the study period.
Hawthorne effect - Mood status | 1-week
  It will be measure if the data collection method affects mood status, by comparing mood status at baseline with results collected over the study period ("Circumplex Mood Model" scale).
Agreement of information (mobile app vs. questionnaire on mood status) | 4-weeks
  It will be assessed in the intervention arm, by comparing the results obtained from the mobile app with those obtained from the self-reported data collected by the "Circumplex Mood Model" scale.
Agreement of information (mobile app vs. questionnaire on physical activity) | 4-weeks
  It will be assessed in the intervention arm, by comparing the results obtained from the mobile app with those obtained from the self-reported data collected by IPAQ-S questionnaire.
Preference of methods | 4-weeks
  Participants of both arms will answer the following question: "If you could choose to participate through an app that measures your movements and asks you to fill in your emotions daily, or through short weekly online/mailed questionnaires, what would you choose? Why?"

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Barros, Professor, Principal Investigator — Institute of Public Health of the University of Porto (ISPUP)